# The effect of different altitude levels on spinal anesthesia in cesarean section surgery; Comparison of anesthesia parameters and hemodynamic changes

| DEMOGRAPHIC DA | ATA; | | | | | | | | <br> |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | <br> |
| Age | | | | | | | | | |
| Weight/Height/<br>BMI | | | | | | | | | |
| (m-kg-kg/m2) | | | | | | | | | |
| ASA | | | | | | | | | |
| INTRAOPERATIVE | FOLLOW | ′-UP; | | | | | | | |
| | Basal | After<br>Spinal<br>3.minute | 5.mn | 10.mn | 15.mn | 30.mn | 45.mn | 60.m<br>n | |
| HR (Heart rate) | | | | | | | | | |
| MAP (mean<br>arterial pressure)<br>mmHg | | | | | | | | | |
| SpO2(Saturation) | | | | | | | | | |
| Number and du | ration | of spinal a | nesthes | sia | | | | | |
| applications | | | | | | | | | |
| The value meas | sured w | rith a pH n | neter | | | | | | |
| Sensory block T6 | transit | time | | | | | | | |
| Highest level of s | sensory | block | | | | | | | |
| MB (modified br | omage) | scale; time | e to read | ch score | 1 | | | | |

| MB (modified bromage) scale; time to reach score 2 |
|----------------------------------------------------|
| MB (modified bromage) scale; time to reach score 3 |
| Number of hypotensive episodes requiring |
| ephedrine |
| Number of episodes of bradycardia requiring |
| atropine |
| Number of episodes of nausea requiring Zofer |
| Surgery time |
| Anesthetic complications |

#### POSTOPERATIF TAKIP;

| | 1.hour | 2.hour | 3.hour | 4.hour | 5.hour |
|---------------------------|--------|--------|--------|--------|--------|
| Sensory blockade end time | | | | | |
| Motor blockade end time | | | | | |
| Nausea-vomiting | | | | | |

## Postdural puncture headache follow-up (YES/NO)

| 1.day | 7.day |
|-------|-------|

### Modified bromage scale

| 0 | No paralysis, the patient can fully flex the foot and knee |
|---|---------------------------------------------------------------------|
| 1 | Can only move knee and feet, can't lift leg straight |
| 2 | Can't flex knee, can only move foot |
| 3 | He cannot move his foot joint or big toe, he has complete paralysis |

## Nausea-vomiting 'Verbal Descriptive Scale'

| 1: | Mild nausea |
|----|-------------------|
| 2: | Moderate nausea |
| 3: | One time vomiting |
| 4: | Multiple vomiting |

#### Study design

Standard noninvasive blood pressure, heart rate (HR), electrocardiogram (ECG) findings, peripheral oxygen saturation (SpO2) will be monitored for all patients brought to the operating room. 2.2 cc of bupivacaine will be administered after entering the L4-5 space under sterile conditions in the sitting position and seeing the cerebrospinal fluid flow. The shastaol will be quickly tilted laterally. Sensory block level will be checked with pinprick test and surgery will be started by recording the time to reach T6 dermatome. Mean arterial pressure, heart rate and peripheral oxygen saturation will be recorded before the procedure (baseline), at the 3rd, 5th, 10th, 15th, 30th, 45th and 60th minutes after the procedure. The number and duration of spinal anesthesia applications, the duration of sensory block formation in the T6 dermatome, the time to reach each score of the Modified bromage score scale, the operation time (the time from the beginning of the surgical incision to the completion of the surgery), the highest level of sensory block, and anesthetic complications will be recorded. Patients with a sensory block level below T6 in the recovery room and a Modified Aldrete score above 8 will be taken to the ward. During the postoperative period, sensory blockade time (time to feel the S2 dermatome), motor blockade time (time to have a MB score of 0) will be recorded every hour in the ward. Nausea and vomiting in the postoperative period will be followed up with the Verbal Descriptive Scale. On the first and seventh days after the operation, the patients will be questioned by the researcher for postdural puncture headache (PDPH, increased pain intensity when standing up from the supine position) by phone call.